CLINICAL TRIAL: NCT07305168
Title: A Multicenter Retrospective Analysis of Postoperative Respiratory Complications in Children With Obstructive Sleepapnea
Acronym: MRA PORC
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, Vera Saldien, Principal Investigator, University Hospital, Antwerp
Other Study IDs: EDGE 004218
Record Dates: First submitted 2025-11-17; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Obstructive Sleep Apnea; Postoperative Respiratory Complications; Adenotonsillectomy; Child Obesity; Craniofacial Abnormalities; Children With Down Syndrome; Neurologic Disorder
MeSH Terms: conditions — Sleep Apnea, Obstructive; Pediatric Obesity; Craniofacial Abnormalities; Nervous System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children with Obstructive Sleepapnea (OSA): Children with OSA after (adeno)tonsillectomy

SUMMARY:
This retrospective observational study aims to evaluate postoperative respiratory complications (PORC) after (adeno)tonsillectomy in children with OSA.

In order to increase the number of patients available for analysis, we will merge data collected at UZA with data collected at the the Department of Sleep Laboratory and Sleep Surgery at the Heim Pal National Pediatric Institute, Hungary. These colleagues performed an identical prospective data collection.

DETAILED DESCRIPTION:
This is a retrospective, multicenter cohort study using anonymized electronic health record data collected in a prospective study (PORC -EDGE 2364) performed at UZA and an identical prospective data collection performed by collegues at Department of Sleep Laboratory and Sleep surgery at Heim Pal National Pediatric Institute at Budapest.Data are collected from otherwise healthy children and children with varying comorbidities undergoing (adeno)-tonsillecty for Obstructive Sleepapnea (OSAS). Per-postoperative management was carried out according to a predefined treatment protocol.

As this study uses existing data, no informed consent was required. The aim of the current project is to answer the following questions.

* What is the prevalence of Postoperative Respiratory Complications (PORC) in children undergoing surgical treatment for OSA and is the prevalence different according to the underlying comorbid condition (i.e obesity, craniofacial malformation, syndromes Down syndrome, neurological conditions affecting upper airway muscle tone)?
* Which factors are associated with the occurrence of PORC (Polysomnogram (PSG) related factors such as obstructive Apnea-Hypopnea Index (oAHI), minimum oxygen saturation during PSG, and patient related factors such as age at time of surgery, presence of a comorbidity)?
* Is it possible to develop a management algorithm for postoperative management based upon the risk factors for PORC above.

ELIGIBILITY:
Inclusion Criteria:

* scheduled for (adeno)tonsillectomy as treatment for OSAS

Exclusion Criteria:

* other surgery than (adeno)tonsillectomy performed as treatment for OSAS
* Polysomnography not available within 1 year before surgery

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: children with or without co-morbidities undergoing (adeno)tonsillectomy for OSAS during time frame of the study period
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-05-02 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
What is the prevalence of PORC in children undergoing surgical treatment for OSA and is the prevalence different according to the underlying comorbid condition | 24 hours postoperative
  Number of PORC

CONTACTS AND LOCATIONS:
Overall Officials: Vera Saldien, MD, Principal Investigator — University Hospital, Antwerp
Locations (2):
- Antwerp University Hospital, Edegem, Antwerp, Belgium
- Heim Pal Children's Hospital, Budapest, Hungary